CLINICAL TRIAL: NCT01766388
Title: Mifepristone and Misoprostol for Mid-trimester Termination of Pregnancy (13-22 Weeks LMP) in Armenia
Brief Title: Mifepristone and Misoprostol for Mid-trimester Termination of Pregnancy in Armenia
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1005
Record Dates: First submitted 2012-12-06; First posted 2013-01-11 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Abortion in Second Trimester

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women of 13-22 weeks gestation

SUMMARY:
The primary goal of this study is to examine the efficacy and feasibility of a mifepristone combined with misoprostol medical abortion regimen in terminating pregnancies 13-22 weeks in Armenia.

DETAILED DESCRIPTION:
Women who were deemed eligible for the study by the provider gave informed consent. They took 200 mg of mifepristone orally at the study clinic. In 24-44 hours, they returned to the clinic for induction with misoprostol. They were admitted as inpatients at the clinic and took 400 mcg of buccal misoprostol every 3 hours until the fetus and placenta were expelled. If there was no full expulsion after 10 doses of misoprostol, the provider used their discretion to determine the appropriate clinical course of action. After responding to questions about their experience with the procedure, women were discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy of 13-22 weeks' gestation
* Good general health
* Meeting legal criteria to obtain abortion
* Presenting with closed cervical os and no vaginal bleeding
* Live fetus at time of presentation for service
* Willingness to undergo a surgical completion if necessary
* No contraindications to study procedures, according to provider
* Woman willing and able to consent to procedure, either by reading consent document or by having consent document read to her
* Willingness to follow study procedures

Exclusion Criteria:

* Known previous transmural uterine incision
* Known allergy to mifepristone or misoprostol/prostaglandin or other contraindications to the use of mifepristone or misoprostol
* Parity greater than 5
* Any contraindications to vaginal delivery, including placenta previa
* Presentation in active labor (defined as moderate to severe contractions every 10 minutes or less)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women presenting to a study clinic in Yerevan, Armenia for voluntary termination of intrauterine pregnancy with gestational ages of 13-22 weeks
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Rate of successful abortion | Every 3 hours after induction with misoprostol commences, up to 30 hours after the first dose

SECONDARY OUTCOMES:
Total dose of misoprostol | At the time of fetal and placental expulsion, up to 30 hours after the first dose
Women's satisfaction with the method | At discharge, up to 5 days after enrollment
Side effects | Every 3 hours, starting from the first dose of misoprostol, up to fetal and placental expulsion or 30 hours after the first dose, whichever occurs first
Women's acceptability of the side effects, buccal administration of misoprostol, and duration of procedure | At discharge, up to 5 days after enrollment
Providers' acceptability of the method | After all study procedures complete, at close out, up to 1.5 years after study enrollment commences
Complications including heavy bleeding, uterine rupture, or infection requiring additional treatment | Every 3 hours, starting from the first dose of misoprostol, up to fetal and placental expulsion, or 30 hours after the first dose, whichever occurs first
Induction to fetal expulsion interval | Time from administration of first misoprostol dose to expulsion of the fetus, up to 30 hours after the first dose
Induction to fetal and placental expulsion interval | Time from administration of first misoprostol dose to expulsion of the fetus and placenta, up to 30 hours after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Ruzanna Abrahamyan, MD, Principal Investigator — Republican Institute of Reproductive Health, Perinatology, Obstetrics and Gynecology; Gayane Abrahamyan, MD, PhD, Principal Investigator — State Medical University; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (2):
- Armenia (2):
  - State Medical University, Yerevan
  - Republican Institute of Reproductive Health, Perinatology, Obstetrics and Gynecology, Yerevan